CLINICAL TRIAL: NCT02188680
Title: Does Irritable Bowel Syndrome Improved by Low FODMAP Diet ?
Brief Title: Irritable Bowel Syndrome and Low FODMAP Diet
Acronym: FructIBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/011/HP
Record Dates: First submitted 2013-08-26; First posted 2014-07-11 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2023-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: fructose test
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low FODMAPS diet and positive breath testing for fructose (Active Comparator): Patients with breath testing positive have a low FODMAPS diet. The test will be considered as positive if we observe an increase of more than 20 ppm of H2 and/or CH4 on a sample with regard to the basal concentration
  Interventions: Other: Low FODMAPS diet
- negative breath testing for fructose (Sham Comparator): patients with negative breath test have a low FODMAPS diet
  Interventions: Other: Low FODMAPS diet

INTERVENTIONS:
Other: Low FODMAPS diet — FODMPAS low diet in patients with IBS and positive breath test for fructose FODMAPS low diet in patients with IBS and negative breath test for fructose

SUMMARY:
The patients having a syndrome SII would be more intolerant in the fructose than the healthy subjects and would benefit from a fructose diet but also from the fructans which contain some fructose. The intolerance in the fructose is diagnosed thanks to a respiratory test after absorption of fructose. However, the eviction of the fructose is sometimes recommended to the patients without having realized beforehand the test of intolerance.

DETAILED DESCRIPTION:
The main objective is to evaluate the efficacy of the FODMAPS diet on IBS symptoms and to correlate the results with the respiratory test

ELIGIBILITY:
Inclusion Criteria:

* older than 18, patients with IBS, patients with no organic disorders, patients informed and agreed to participate

Exclusion Criteria:

* patients with sclerodermia, diabetes, obesity, anorexia, colo-rectal surgery, patients with small intestinal bacterial overgrowth, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Fructose expiration rate (ppm) | Day 15
  Estimate the value of the fructose test to predict the efficiency of a diet excluding the fructose and its by-products on the digestive symptoms of the patients having a Syndrome of the irritable bowel.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie LEROI, Professor, Principal Investigator — University Hospital, Rouen
Locations (1):
- Service de Physiologie Digestive, Urinaire, Respiratoire et Sportive, Rouen, Haute Normandie, France

REFERENCES:
- [Derived] Melchior C, Desprez C, Houivet E, Debeir LA, Bril L, Maccarone M, Grout E, Ducrotte P, Gourcerol G, Leroi AM. Is abnormal 25 g fructose breath test a predictor of symptomatic response to a low fructose diet in irritable bowel syndrome? Clin Nutr. 2020 Apr;39(4):1155-1160. doi: 10.1016/j.clnu.2019.04.031. Epub 2019 May 8. PMID 31113646